CLINICAL TRIAL: NCT05960929
Title: InfasurfAero™ Versus Sham Treatment in Preterm Newborns With RDS: A Single-dose, Double-blind, Random Allocation, Sham-control, Clinical Trial
Brief Title: InfasurfAero™ Versus Sham Treatment in Preterm Newborns With RDS
Acronym: Aero-05
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ONY (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AERO-05 Protocol
Record Dates: First submitted 2023-07-06; First posted 2023-07-27 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-11

CONDITIONS: Respiratory Distress Syndrome (Neonatal); Intubation Complication; Death; Neonatal
Keywords: Infasurf; Calfactant; Inhalation; Nebulization; Preterm; InfasurfAero; Respiratory Distress Syndrome; Neonatal; NICU; CPAP; Intubation; Aerosol; CPAP Failure
MeSH Terms: conditions — Pulmonary Atelectasis; Perinatal Death; Respiratory Aspiration; Premature Birth; Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: This single-dose, double-blind, random allocation, sham-control, clinical trial will recruit spontaneously breathing newborns with RDS stable on non-invasive nasal respiratory support. Enrolled clinical study subjects will be randomly allocated to receive respiratory air with Infasurf® (Intervention Arm) or respiratory air alone (Sham Control Arm) through the InfasurfAero™.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All study procedures will be performed behind a portable screen or curtain, or in a separate procedure room so that non-study personnel (including the primary care team) will be unaware of the subject's assigned study arm. Study personnel involved in the study procedure will not be masked. All other study personnel including the investigator and the outcomes accessor will be masked throughout the duration of the study.
  The subject's family will remain blinded to treatment assignment throughout.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment Arm (Experimental): A single dose of Calfactant at 6ml/kg administered via the Infasurf Aero™ Nebulizer until completion.
  Interventions: Combination Product: Infasurf Aero™
- Control Arm (Sham Comparator): Low flow respiratory air alone through the InfasurfAero™ Nebulizer until completion.
  Interventions: Combination Product: Infasurf Aero™

INTERVENTIONS:
Combination Product: Infasurf Aero™ — A single dose of Calfactant administered by pacifier interface by inhalation via the Infasurf Aero nebulizer at 6ml/kg.

SUMMARY:
The purpose of this clinical study is to determine the effectiveness and safety of Infasurf® administered through the InfasurfAero™, a novel oral airway delivery device specifically designed to give Infasurf in a less complicated way and without the need for a breathing tube or interrupting nasal respiratory support.

DETAILED DESCRIPTION:
This single-dose, double-blind, random allocation, sham-control, clinical trial will recruit spontaneously breathing newborns with RDS stable on non-invasive nasal respiratory support. Enrolled clinical study subjects will be randomly allocated to receive respiratory air with Infasurf® (Intervention Arm) or respiratory air alone (Sham Control Arm) through the InfasurfAero™.

The objectives of this clinical study are to i) assess the effectiveness of a single dose of Infasurf administered through the InfasurfAero in preventing CPAP failure, and ii) assess the safety of Infasurf administered through the InfasurfAero.

Subjects will be enrolled at one of 10+ sites. 7 sites are currently recruited.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria include ALL of the following:

1. Written informed consent obtained by parent or legal representative prior to or after birth
2. Gestational age at birth ≥ 29 0/7 AND ≤ 35 6/7 weeks
3. Birthweight ≥ 1,000 AND ≤ 3,500 grams
4. Age ≥ 1 hour AND ≤ 6 hours
5. Clinical diagnosis of surfactant-deficient RDS, with EITHER i. a Silverman-Anderson Retraction Score ≥ 5 (in Room Air), OR ii. signs of respiratory distress (tachypnea, retractions, grunting) AND radiographic confirmation
6. Require CPAP
7. Respiratory Severity Score (RSS) ≥ 1.25 AND ≤ 2.4
8. If subject is >346/7 weeks' gestation a chest radiograph is required

Exclusion Criteria:

Exclusion criteria are ANY of the following:

1. Surfactant administration prior to randomization
2. Mechanical ventilation prior to randomization
3. Major congenital anomaly (suspected or confirmed)
4. Abnormality of the airway (suspected or confirmed)
5. Respiratory distress presumed secondary to an etiology other than RDS (e.g., suspected pulmonary hypoplasia, pneumothorax, meconium aspiration syndrome, pneumonia, septic or hypovolemia shock, hypoxic ischemic encephalopathy)
6. Apgar score < 3 at 5 minutes of age
7. Umbilical cord gas pH <7.0 or BD > 10
8. Any condition that, in the opinion of the Investigator, would place the neonate at undue risk

Ages: 29 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
CPAP failure and or death | Within 1st week of age
  CPAP failure is defined as a respiratory severity score (RSS) (MAP x FiO2) >2.5 on two consecutive assessments at least 30 minutes apart, or an RSS > 2.4 and one or more of the following:
  (i) Silverman-Andersen respiratory severity score (https://www.thecalculator.co/health/Silverman-Score-Calculator-1125.html) of ≥ 5 despite respiratory support.
  (ii) Severe apnea (2 or more episodes per hour, or 1 or more episodes requiring manual positive pressure ventilation).
  (iii) Respiratory acidosis (pCO2 > 65 with a pH < 7.2 on blood gas). RSS will be the primary indicator of CPAP failure. However with the addition of the Silverman-Anderson scores, severe apnea and respiratory acidosis, CPAP failure may occur earlier than solely defined by RSS score.

SECONDARY OUTCOMES:
Chronic lung disease and or death | 36 weeks post menstrual age (PMA).
  Chronic lung disease is defined as altitude adjusted oxygen requirement at 36 weeks post menstrual age.
Incidence of MV | 36 weeks PMA
  Incidence of Mechanical Ventilation
Duration of MV | 36 weeks PMA
  length of time of Mechanical Ventilation
Incidence of intubation | 36 weeks PMA
  Any occurrence of tracheal intubation
Incidence of invasive surfactant replacement therapy | 72 hours post birth
  any occurrence of liquid surfactant administration via and endotracheal tube
Duration of non-invasive support | 36 weeks PMA
  Length of time of respiratory support other than Intubation
Duration of supplemental oxygen | 36 weeks PMA
  Length of time any oxygen is administered.

OTHER OUTCOMES:
Adverse events during surfactant administration. | Birth to 72 hours of age.
  Incidence of bradycardia and desaturation during surfactant administration.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Guthrie, MD, Study Chair — Vanderbilt Jackson-Madison, Jackson TN; Dinushan Kaluarachchi, MD, Study Chair — Unity Point Meriter, Madison WI; Jim Cummings, MD, Study Director — Ony Biotech
Locations (10):
- United States (10):
  - St. Josephs Hospital and Medical Center, Phoenix, Arizona
  - Phoenix Children's, Phoenix, Arizona
  - Sharp Mary Birch Hospital for Women & Newborns, San Diego, California
  - University of Florida -Jacksonville, Jacksonville, Florida
  - Kapi'olani Medical Center for Women & Children, Honolulu, Hawaii
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Sisters of Charity Hospital, Buffalo, New York
  - Western TN- Jackson-Madison County General Hospital, Jackson, Tennessee
  - Utah Valley Hospital, Provo, Utah
  - Unity Point Meriter, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No